CLINICAL TRIAL: NCT02062853
Title: CQI Pilot Study Evaluating the Utility of an Educational Video in the Setting of Topical 5-fluorouracil Therapy to Treat Actinic Keratoses and Its Influence on Patient Satisfaction
Brief Title: Continuous Quality Improvement (CQI) Pilot Study Evaluating the Utility of an Educational Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 384968; 384968 (Other: University of California, Davis)
Record Dates: First submitted 2013-11-26; First posted 2014-02-14 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Group (Experimental): Subjects view educational video on the use of cream medication for the treatment of actinic keratoses.
  Interventions: Other: Video Group
- Verbal Group (Active Comparator): Subjects are given verbal instructions on the use of cream medication for the treatment of actinic keratoses.
  Interventions: Other: Verbal Group

INTERVENTIONS:
Other: Video Group — Subjects will view a brief video today (about 5 minutes long) that provides information on the cream medication that will be used for treatment of your actinic keratoses.
  Arms: Video Group
Other: Verbal Group — The physician will provide information about the cream medication for the treatment of actinic keratoses through a regular conversation.
  Arms: Verbal Group

SUMMARY:
The primary aim of this study is to evaluate the effects of prospective patient education on patient satisfaction with administration of topical 5% 5-fluorouracil cream for the treatment of actinic keratosis involving the face, scalp, upper chest, dorsal hands and forearms. Specifically, this study aims to determine if prospective patient viewing of an educational video delineating treatment effects and expectations improves patient satisfaction and treatment completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of actinic keratoses with at least 6 clinically-diagnosed actinic keratoses on the face, bald scalp, arms, upper chest, OR dorsal hands classified as grade I, mild (slightly palpable actinic keratoses, more easily felt than seen), and II, moderate (moderately thick hyperkeratotic actinic keratoses, easily felt).

Exclusion Criteria:

* Patients using interferon or interferon inducers, immunomodulators, cytotoxic or immunosuppressor drugs, corticosteroids, retinoids, or investigational drugs within 4 weeks prior to enrollment.
* Patients who have been treated with any topical drug for actinic keratoses lesions less than 8 weeks prior to enrollment.
* Patients with invasive tumors within the treated area (e.g. invasive squamous cell carcinoma)
* Patients who have exhibited any dermatological disease within the treated or adjacent (3 cm distance) area at the time of screening.
* Patients who have known allergies to fluorouracil (5-FU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Level of Patient Satisfaction in Relation to Treatment Effects and Expectations of 5-fluorouracil Cream | 4 weeks
  The level of patient satisfaction will be assessed via questionnaire and visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Fazel, M.D., D.D.S., Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical